CLINICAL TRIAL: NCT04110366
Title: Kinetics of Mucosal and Systemic Immune Responses to Intranasal Live Attenuated Influenza Vaccine (LAIV)
Brief Title: Nasal and Systemic Immune Responses to Nasal Influenza Vaccine
Acronym: Flu-M3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18/LO/0904
Record Dates: First submitted 2019-09-09; First posted 2019-10-01 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Influenza; Vaccine Virus Shedding
Keywords: influenza; vaccine; virus; antibody; cytokine; respiratory
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live attenuated influenza vaccine (Experimental): Participants receiving live attenuated influenza vaccine (LAIV)
  Interventions: Biological: Live attenuated influenza vaccine
- Mucosal immune stability cohort (Experimental): Participants receiving a vehicle control nasal challenge
  Interventions: Other: Vehicle control

INTERVENTIONS:
Biological: Live attenuated influenza vaccine — Vaccination with live attenuated influenza vaccine (LAIV)
  Other Names: Fluenz
  Arms: Live attenuated influenza vaccine
Other: Vehicle control — Vehicle control nasal challenge
  Arms: Mucosal immune stability cohort

SUMMARY:
Intranasal live attenuated influenza vaccine (LAIV; trade name FluMist/Fluenz-Tetra, manufactured by AstraZeneca/Medimmune) is the standard influenza vaccine given to children aged 2-17 years of age in the UK. It is also licensed to be given to adults up to the age of 49 years in the USA. The systems biology of the human blood response to influenza vaccines has been studied in great detail, but there is a paramount need to study innate and specific, soluble and cellular immune responses at the nasal mucosal site of influenza infection. In this way this study aims to determine correlates of efficacy and vaccine take in serum and nasal mucosal lining fluid (MLF).

DETAILED DESCRIPTION:
This study will collect serial samples prior to vaccination and at intervals up to day 28 post-vaccination to establish the kinetics of the nasal mucosal and blood systemic response to LAIV in young adults aged 18-30 years (n=40). In the nose the investigators will measure viral load, soluble mediators of inflammation and antibodies (humoral immunity) in mucosal lining fluid; while cellular immune responses and serology will be assessed in blood samples. Investigators at Imperial College London (ICL) have been involved in the development of novel methods of non-invasive precision mucosal sampling, including absorption of MLF from the nose by nasosorption. The investigators have also developed assays for influenza-specific IgA by ELISA, and aim to compare this assay against a repertoire of serological assays in patients after LAIV administration.

The study will precisely assess mucosal and systemic immune responses to the LAIV nasal vaccine.

The primary endpoint will be based on nasal mucosal levels of IgA and IgG antibodies to the 4 constituent viral subtypes in LAIV: measured by ELISA and multiplex immunoassay (Mesoscale Diagnostics) and expressed as seroconversion rates, geometric mean titre (GMT) changes, and geometric mean fold rises (GMFR). The secondary endpoints will be: (1) haemagglutination inhibition (HAI) assay titres measured in serum and the nose, (2) influenza pseudotype neutralisation by antibodies in serum and the nose, (3) nasal cytokine and chemokine levels as measured by immunoassay and (4) nasal viral load quantified by qPCR.

It is thought that the immune response to LAIV in an individual is mediated by a combination of mucosal and systemic factors, involving innate and specific mechanisms that have different kinetics, and various cell types. By understanding the molecular and cellular basis of the nasal mucosal response to LAIV, the investigators hope to identify key molecular signatures and biomarkers associated with LAIV responses, and to assess protective pathways that could be stimulated by novel vaccines. The nasal vaccine challenge model could be used to test other new vaccines, and proceed to rational development of improved vaccines for influenza and other diseases. Furthermore nasal mucosal methods could be used in the clinic to identify subjects who have responded poorly to vaccines, or to assess vaccine efficacy in large populations.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide written informed consent
* Aged 18-30 years (inclusive)
* Fluent English speaker

Exclusion Criteria:

* Current involvement in another study unless observational or in follow-up phase (non-interventional)
* Received any influenza vaccine over the last 2 years
* Egg allergy
* Previous significant adverse reaction to any vaccination/immunisation
* Current regular (daily) smoker
* Pregnant
* Any medication that may affect the immune system (e.g. steroids)
* Taking regular acetylsalicylic acid (aspirin)
* Unable to give informed consent
* Current acute severe febrile illness
* Taking long term antibiotics
* Clinically diagnosed influenza in the last 2 years
* Any long-term health problem with heart disease, lung disease (including asthma), kidney disease, neurologic disease, liver disease, metabolic disease (e.g. diabetes) or anemia or another blood disorder
* Use of drugs for the treatment of rheumatoid arthritis, Crohn's disease, or psoriasis or anticancer drugs; or radiation treatments
* History of Guillain-Barre syndrome
* Live with or expect to have close contact with a person whose immune system is severely compromised and who must be in protective isolation (e.g., an isolation room of a bone marrow transplant unit)
* Received any other vaccinations in the past 4 weeks

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Openshaw, PhD, Principal Investigator — Imperial College London; Trevor T Hansel, PhD, Study Director — Imperial College London
Locations (1):
- Imperial Clinical Respiratory Research Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing is available upon request to the study PI; but access is offered at the discretion of the PI and requests are not guaranteed access. All access will require ethical approval.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: From June 2020 onward, no set end date
Access Criteria: PI discretion

REFERENCES:
- [Derived] Thwaites RS, Uruchurtu ASS, Negri VA, Cole ME, Singh N, Poshai N, Jackson D, Hoschler K, Baker T, Scott IC, Ros XR, Cohen ES, Zambon M, Pollock KM, Hansel TT, Openshaw PJM. Early mucosal events promote distinct mucosal and systemic antibody responses to live attenuated influenza vaccine. Nat Commun. 2023 Dec 5;14(1):8053. doi: 10.1038/s41467-023-43842-7. PMID 38052824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events occur after participant enrollment but prior to assignment to a study arm. Participants were not randomised for assignment to LAIV or Mucosal immune stability arms, but were assigned based on their having responded to different enrollment advertisements.
Groups:
- Live Attenuated Influenza Vaccine: Participants receiving live attenuated influenza vaccine (LAIV) were initially screened per the study protocol to ensure that inclusion and exclusion criteria were complete. Participants were then invited to the vaccination arm of the study, where n=40 participants received LAIV and completed 5 study visits each over the course of 28 days.
- Mucosal Immune Stability Cohort: Vehicle control nasal challenge recipients n=8
Period: Overall Study
Arm/Group | Live Attenuated Influenza Vaccine | Mucosal Immune Stability Cohort
Started | 40 | 8
Completed | 40 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population does not differ from the Participant Flow.
Groups:
- Mucosal Immune Stability Cohort: In the placebo/vehicle challenge 'Mucosal immune stability' arm, a further n=8 participants attended for a single visit at which repeat nasal samples were collected to match the LAIV arm.
- Total: Total of all reporting groups
Arm/Group | Live Attenuated Influenza Vaccine | Mucosal Immune Stability Cohort | Total
Number analyzed (Participants) | 40 | 8 | 48
Age, Continuous [Median (Full Range); unit: years] | 22 [18 to 29] | 23 [18 to 25] | 22 [18 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 5 | 35
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 8 | 48
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Shedding Each Vaccine Virus Measured by qPCR of Nasosorption Samples
Description: Vaccine virus shedding in nasosorption samples collected between 1-7 days post-vaccination and quantified using multiplex qPCR assay measures in the LAIV vaccine recipient cohort.
Time Frame: 1-7 days post vaccination
Population: All participants
Measure: Number; unit: participants
Groups:
- Live Attenuated Influenza Vaccine: Participants receiving live attenuated influenza vaccine (LAIV) were initially screened per the study protocol to ensure that inclusion and exclusion criteria were complete. Participants were then invited to the vaccination arm of the study, where n=40 participants received LAIV and completed 5 study visits each over the course of 28 days.
  n=31 participants (78%) shed at least one vaccine virus, measured by qPCR, on at least one study timepoint.
- Mucosal Immune Stability Cohort: Stability of cytokine levels measured in nasosorption samples collected from participants for the 8 hour duration of this arm. Cytokines measured by multiplex immunoassays.
Arm/Group | Live Attenuated Influenza Vaccine | Mucosal Immune Stability Cohort
Number analyzed (Participants) | 40 | 0
participants | 31 |

2. Secondary Outcome: Number of Participants With >2-fold Rise in Mucosal and/or Serum Antibody Titre Against Each Vaccine Virus Haemagglutinin Antigens
Description: Vaccine specific antibody (IgG and IgA) titres in serum and/or respiratory secretions (nasosorption and nasal wash) measured using endpoint titre and arbitrary unit level immunoassay measurements of samples collected from the n=40 LAIV vaccine recipient arm.
Time Frame: 28 days post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Influenza Vaccine
Number analyzed (Participants) | 40
Participants | 28

ADVERSE EVENTS:
Time Frame: 1 month study duration for vaccine arm, 1 day for placebo control arm.
Groups:
- Mucosal Immune Stability Cohort: In the placebo/vehicle challenge 'Mucosal immune stability' arm, a further n=8 participants attended for a single 8 hour visit at which repeat nasal samples were collected to match the LAIV arm.
Arm/Group | Live Attenuated Influenza Vaccine | Mucosal Immune Stability Cohort
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/8
Other Adverse Events (participants affected / at risk) | 0/40 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04110366/Prot_SAP_000.pdf